CLINICAL TRIAL: NCT00483756
Title: A Phase 2 Randomized, Multicenter, Active Comparator-Controlled Trial to Evaluate the Safety and Efficacy of Co-administration of CP-690,550 and Mycophenolate Mofetil / Mycophenolate Sodium in De Novo Renal Allograft Recipients
Brief Title: Study of a JAK3 Inhibitor for the Prevention of Acute Rejection in Kidney Transplant Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: A3921030
Record Dates: First submitted 2007-06-06; First posted 2007-06-07 (Estimated); Results first posted 2013-03-14 (Estimated); Last update posted 2013-03-14 (Estimated); Status verified 2013-02

CONDITIONS: Kidney Transplantation
Keywords: Immunosuppression; JAK3 inhibitor; kidney transplantation.
MeSH Terms: interventions — Cyclosporine; tofacitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Active Comparator): Treatment Arm 1 will also receive standard of care medications
  Interventions: Drug: Cyclosporine
- 2 (Experimental): Treatment Arm 2 will also receive standard of care medications
  Interventions: Drug: CP-690,550
- 3 (Experimental): Treatment Arm 3 will also receive standard of care medications
  Interventions: Drug: CP-690,550

INTERVENTIONS:
Drug: Cyclosporine — Standard of care
  Arms: 1
Drug: CP-690,550 — CP-690,550 15 mg BID for Months 1-6, then 10 mg BID for Months 7-12
  Arms: 2
Drug: CP-690,550 — CP-690,550 15 mg BID for Months 1-3, then 10 mg BID for Months 4-12
  Arms: 3

SUMMARY:
A new immunosuppressive drug, based on the inhibition of an important enzyme in the immune system called JAK3, is being developed by Pfizer to prevent transplant rejection. In this research study, a JAK3 inhibitor or cyclosporine will be given to new kidney transplant patients for 12 months. Patients will be assigned to one of three treatment groups after receiving a kidney transplant. Two of the treatment groups will receive 2 different dosing regimens of the JAK3 inhibitor that will be taken by mouth. The third treatment group will be a standard-of-care control arm. Patients will continue to take the assigned study medication for 12 months as well as other standard transplant medications such as prednisone.

ELIGIBILITY:
Inclusion Criteria:

* Recipient of a first-time kidney transplant
* Between the ages of 18 and 70 years, inclusive

Exclusion Criteria:

* Recipient of any non-kidney transplant

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 338 (Actual)
Dates: Start 2007-08; Primary Completion 2010-02 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (57):
- United States (28):
  - Pfizer Investigational Site, Little Rock, Arkansas
  - Pfizer Investigational Site, Los Angeles, California
  - Pfizer Investigational Site, Palo Alto, California
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, San Francisco, California
  - Pfizer Investigational Site, Stanford, California
  - Pfizer Investigational Site, Aurora, Colorado
  - Pfizer Investigational Site, New Haven, Connecticut
  - Pfizer Investigational Site, Gainesville, Florida
  - Pfizer Investigational Site, Gainsville, Florida
  - Pfizer Investigational Site, Tampa, Florida
  - Pfizer Investigational Site, Chicago, Illinois
  - Pfizer Investigational Site, Baltimore, Maryland
  - Pfizer Investigational Site, Boston, Massachusetts
  - Pfizer Investigational Site, Springfield, Massachusetts
  - Pfizer Investigational Site, Ann Arbor, Michigan
  - Pfizer Investigational Site, Detroit, Michigan
  - Pfizer Investigational Site, Rochester, Minnesota
  - Pfizer Investigational Site, St Louis, Missouri
  - Pfizer Investigational Site, Livingston, New Jersey
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Valhalla, New York
  - Pfizer Investigational Site, Chapel Hill, North Carolina
  - Pfizer Investigational Site, Portland, Oregon
  - Pfizer Investigational Site, Philadelphia, Pennsylvania
  - Pfizer Investigational Site, Charleston, South Carolina
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, Fort Worth, Texas
- Australia (6):
  - Pfizer Investigational Site, Camperdown, New South Wales
  - Pfizer Investigational Site, Westmead, New South Wales
  - Pfizer Investigational Site, Adelaide, South Australia
  - Pfizer Investigational Site, Woodville, South Australia
  - Pfizer Investigational Site, Clayton, Victoria
  - Pfizer Investigational Site, Parkville, Victoria
- Belgium (2):
  - Pfizer Investigational Site, Anderlecht
  - Pfizer Investigational Site, Leuven
- Brazil (2):
  - Pfizer Investigational Site, Porto Alegre, Rio Grande do Sul
  - Pfizer Investigational Site, São Paulo, São Paulo
- Pfizer Investigational Site, Edmonton, Alberta, Canada
- Pfizer Investigational Site, Prague, Czechia
- France (4):
  - Pfizer Investigational Site, Nantes
  - Pfizer Investigational Site, Paris
  - Pfizer Investigational Site, Toulouse
  - Pfizer Investigational Site, Vandœuvre-lès-Nancy
- Germany (2):
  - Pfizer Investigational Site, Berlin
  - Pfizer Investigational Site, Hamburg
- Italy (2):
  - Pfizer Investigational Site, Bologna
  - Pfizer Investigational Site, Roma
- Pfizer Investigational Site, Rotterdam, Netherlands
- Pfizer Investigational Site, Oslo, Norway
- Poland (2):
  - Pfizer Investigational Site, Warsaw
  - Pfizer Investigational Site, Wroclaw
- Portugal (2):
  - Pfizer Investigational Site, Coimbra
  - Pfizer Investigational Site, Lisbon
- Pfizer Investigational Site, Seoul, South Korea
- Spain (2):
  - Pfizer Investigational Site, Barcelona, Barcelona
  - Pfizer Investigational Site, L'Hospitalet de Llobregat, Barcelona

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3921030&StudyName=Study%20of%20a%20JAK3%20Inhibitor%20for%20the%20Prevention%20of%20Acute%20Rejection%20in%20Kidney%20Transplant%20Patients

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Initially 7 participants were enrolled and randomized under original protocol but enrollment was terminated because 2 participants developed Grade 2B rejection. Protocol amendment 1 was implemented to increase aggregate level of immunosuppression and 331 participants were enrolled. Results of participants enrolled under amendment 1 are reported.
Groups:
- Cyclosporine: Cyclosporine (CsA) microemulsion at a starting dose of 8 to 10 milligram per kilogram per day (mg/kg/day) orally twice daily in 2 equal doses for 12 months. Dosages were adjusted according to trough whole blood level and standard institutional practice. Participants also received mycophenolate mofetil tablet 1 gram orally twice daily (up to 1.5 gram orally twice daily in Black participants) for 12 months.
- CP-690,550 15 mg for Months 1 to 6: CP-690,550 15 milligram (mg) tablet orally twice daily for Month 1 to 6, then 10 mg tablet orally twice daily for Month 7 to 12. Participants also received mycophenolate mofetil 1 gram tablet orally twice daily for 12 months.
- CP-690,550 15 mg for Months 1 to 3: CP-690,550 15 mg tablet orally twice daily for Month 1 to 3, then 10 mg tablet orally twice daily for Month 4 to 12. Participants also received mycophenolate mofetil 1 gram tablet orally twice daily for 12 months.
Period: Overall Study
Arm/Group | Cyclosporine | CP-690,550 15 mg for Months 1 to 6 | CP-690,550 15 mg for Months 1 to 3
Started | 110 | 110 | 111
Treated | 109 | 106 | 107
Completed | 77 | 60 | 59
Not Completed | 33 | 50 | 52
Not completed — Death | 2 | 0 | 1
Not completed — Adverse Event | 19 | 38 | 40
Not completed — Lack of Efficacy | 1 | 0 | 0
Not completed — Lost to Follow-up | 3 | 1 | 0
Not completed — Withdrawal by Subject | 5 | 3 | 4
Not completed — Other | 2 | 4 | 3
Not completed — Randomized, Not Treated | 1 | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cyclosporine | CP-690,550 15 mg for Months 1 to 6 | CP-690,550 15 mg for Months 1 to 3 | Total
Number analyzed (Participants) | 109 | 106 | 107 | 322
Age, Customized [Number; unit: participants]
  18 to 44 Years | 45 | 43 | 46 | 134
  45 to 64 Years | 57 | 54 | 56 | 167
  Greater Than or Equal to (>=) 65 Years | 7 | 9 | 5 | 21
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 24 | 27 | 90
  Male | 70 | 82 | 80 | 232

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With First Clinical Biopsy Proven Acute Rejection (BPAR) Episode 6 Months Post-Transplant
Description: Clinical BPAR was a BPAR (category acute rejection as interpreted by the central blinded pathologist according to the Banff 97 working classification) associated with an increase in serum creatinine of >= 0.3 milligram per deciliter (mg/dL) and >=20 percent (%) from pre-rejection baseline. The increase in serum creatinine was assessed based on the comparison of baseline and the highest serum creatinine recorded within 24 hours (hrs) of the time of biopsy.
Time Frame: Baseline up to Month 6
Population: Full analysis set (FAS) with last dosing risk set: all randomized participants who received at least 1 dose of study medication, including events occurring up to 7 days after last dose. Here, N (Number of Participants Analyzed) signifies participants evaluable for this measure.
Measure: Number; unit: participants
Arm/Group | Cyclosporine | CP-690,550 15 mg for Months 1 to 6 | CP-690,550 15 mg for Months 1 to 3
Number analyzed (Participants) | 89 | 78 | 74
participants | 9 | 11 | 7

2. Primary Outcome: Glomerular Filtration Rate (GFR) at Month 12
Description: GFR: an index of kidney function. GFR described the flow rate of filtered fluid through the kidney. GFR was calculated using iohexol serum clearance. For determination of iohexol serum clearance, iohexol was administered as an intravenous bolus over 5 minutes immediately after morning dosing of CP-690,550 or CsA on day of GFR evaluation. A normal GFR is greater than (>) 90 milliliter per minute (mL/min), although children and older people usually have a lower GFR. Lower values indicated poor kidney function. A GFR less than (<) 15 mL/min indicated kidney failure.
Time Frame: 2, 3, 4, and 5 hrs post iohexol intravenous bolus at Month 12
Population: FAS: all randomized participants who received at least 1 dose of study medication. Here, N (Number of Participants Analyzed) includes only participants with evaluable data for this measure at Month 12.
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Cyclosporine | CP-690,550 15 mg for Months 1 to 6 | CP-690,550 15 mg for Months 1 to 3
Number analyzed (Participants) | 72 | 56 | 58
mL/min | 54.14 (19.12) | 65.05 (18.81) | 65.37 (20.77)

3. Secondary Outcome: Glomerular Filtration Rate (GFR) at Month 6
Description: GFR: an index of kidney function. GFR described the flow rate of filtered fluid through the kidney. GFR was calculated using iohexol serum clearance. For determination of iohexol serum clearance, iohexol was administered as an intravenous bolus over 5 minutes immediately after morning dosing of CP-690,550 or CsA on day of GFR evaluation. A normal GFR is >90 mL/min, although children and older people usually have a lower GFR. Lower values indicated poor kidney function. A GFR <15 mL/min indicated kidney failure.
Time Frame: 2, 3, 4, and 5 hrs post iohexol intravenous bolus at Month 6
Population: FAS: all randomized participants who received at least 1 dose of study medication. Here, N (Number of Participants Analyzed) includes only participants with evaluable data for this measure at Month 6.
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Cyclosporine | CP-690,550 15 mg for Months 1 to 6 | CP-690,550 15 mg for Months 1 to 3
Number analyzed (Participants) | 80 | 64 | 67
mL/min | 57.29 (18.52) | 67.54 (21.86) | 73.93 (23.72)

4. Secondary Outcome: Number of Participants With Progression of Chronic Allograft Lesions at Month 12
Description: Progression of chronic allograft lesions was defined as an increase in the Banff chronicity score (Banff-CS) in biopsy from the implantation (baseline) biopsy in a given participant. Banff-CS was the sum of the Banff scores for the 4 chronic basic lesions (allograft glomerulopathy [cg] + interstitial fibrosis [ci] + tubular atrophy [ct] + vascular intimal thickening [cv]).The Banff-CS ranged from 0-12, higher score indicated greater lesions and Month 12 Banff-CS greater than the implantation biopsy score indicated progression of lesions.
Time Frame: Month 12
Population: Per protocol (PP) population: all randomized participants who received at least 1 dose of study treatment; excluding participants who had a protocol deviation thought to affect the analyses. Here, N (Number of Participants Analyzed) includes only participants with evaluable data for this measure at both baseline and Month 12.
Measure: Number; unit: participants
Arm/Group | Cyclosporine | CP-690,550 15 mg for Months 1 to 6 | CP-690,550 15 mg for Months 1 to 3
Number analyzed (Participants) | 48 | 46 | 43
participants | 29 | 18 | 19

5. Secondary Outcome: Number of Participants With First Clinical Biopsy Proven Acute Rejection (BPAR) 12 Months Post Transplant
Description: Clinical BPAR was a BPAR (category acute rejection as interpreted by the central blinded pathologist according to the Banff 97 working classification) associated with an increase in serum creatinine of >= 0.3 mg/dL and >=20% from pre-rejection baseline. The increase in serum creatinine was assessed based on the comparison of baseline and the highest serum creatinine recorded within 24 hrs of the time of biopsy.
Time Frame: Baseline up to Month 12
Population: FAS with last dosing risk set: all randomized participants who received at least 1 dose of study medication, including events occurring up to 7 days after last dose. Here, N (Number of Participants Analyzed) signifies participants evaluable for this measure.
Measure: Number; unit: participants
Arm/Group | Cyclosporine | CP-690,550 15 mg for Months 1 to 6 | CP-690,550 15 mg for Months 1 to 3
Number analyzed (Participants) | 83 | 66 | 61
participants | 9 | 11 | 7

6. Secondary Outcome: Number of Participants With Treated Clinical Acute Rejection
Description: Treated clinical acute rejection was defined as an acute rejection episode that was diagnosed based on local biopsy readout and received anti-rejection treatment.
Time Frame: Month 6, 12
Population: FAS with last dosing risk set: all randomized participants who received at least 1 dose of study medication, including events occurring up to 7 days after last dose. Here, N (Number of Participants Analyzed): participants evaluable for this measure; and n: participants who remained at risk at given time point for each group, respectively.
Measure: Number; unit: participants
Arm/Group | Cyclosporine | CP-690,550 15 mg for Months 1 to 6 | CP-690,550 15 mg for Months 1 to 3
Number analyzed (Participants) | 95 | 86 | 80
participants
  Month 6 (n=95,86,80) | 21 | 23 | 18
  Month 12 (n=92,76,69) | 25 | 26 | 18

7. Secondary Outcome: Number of Participants With Combined Banff Rejection Categories (Categories 2, 3, and 4)
Description: Banff 97: standard classification for scoring and classifying rejection of kidney transplant biopsies in 6 diagnostic categories: normal, antibody-mediated rejection, borderline changes: 'suspicious' for acute cellular rejection, acute/active cellular rejection, chronic/sclerosing allograft nephropathy, and other. Combined Banff rejection calculated from categories of antibody-mediated rejection (Category 2) plus borderline changes (Category 3) plus acute rejection (Category 4), as interpreted by the central pathologist.
Time Frame: Month 6, 12
Population: FAS with last dosing risk set: all randomized participants who received at least 1 dose of study medication, including events occurring up to 7 days after last dose. Here, N (Number of Participants Analyzed): participants evaluable for this measure; and n: participants who were evaluable at given time point for each group, respectively.
Measure: Number; unit: participants
Arm/Group | Cyclosporine | CP-690,550 15 mg for Months 1 to 6 | CP-690,550 15 mg for Months 1 to 3
Number analyzed (Participants) | 100 | 83 | 83
participants
  Month 6 (n=100,83,83) | 29 | 22 | 20
  Month 12 (n=96,74,71) | 30 | 24 | 23

8. Secondary Outcome: Number of Participants With Graft Loss
Description: Graft loss was defined as graft nephrectomy, participant death, re-transplantation, or return to dialysis for >=6 consecutive weeks.
Time Frame: Month 6, 12
Population: as for outcome 6
Measure: Number; unit: participants
Arm/Group | Cyclosporine | CP-690,550 15 mg for Months 1 to 6 | CP-690,550 15 mg for Months 1 to 3
Number analyzed (Participants) | 85 | 68 | 72
participants
  Month 6 (n=85,68,72) | 1 | 1 | 3
  Month 12 (n=79,56,58) | 1 | 1 | 3

9. Secondary Outcome: Number of Participants With Efficacy Failure
Description: Efficacy failure was the first occurrence of clinical BPAR diagnosed by the central pathologist or graft loss including participant death.
Time Frame: Month 6, 12
Population: as for outcome 6
Measure: Number; unit: participants
Arm/Group | Cyclosporine | CP-690,550 15 mg for Months 1 to 6 | CP-690,550 15 mg for Months 1 to 3
Number analyzed (Participants) | 98 | 84 | 80
participants
  Month 6 (n=98,84,80) | 21 | 19 | 14
  Month 12 (n=94,74,67) | 22 | 20 | 16

10. Secondary Outcome: Number of Participants Who Died
Time Frame: Month 6, 12
Population: as for outcome 6
Measure: Number; unit: participants
Arm/Group | Cyclosporine | CP-690,550 15 mg for Months 1 to 6 | CP-690,550 15 mg for Months 1 to 3
Number analyzed (Participants) | 86 | 69 | 69
participants
  Month 6 (n=86,69,69) | 2 | 2 | 0
  Month 12 (n=80,57,55) | 2 | 2 | 0

11. Secondary Outcome: Lymphocyte Subset
Description: The absolute cell counts of cluster of differentiation 3 (CD3): T-lymphocytes, cluster of differentiation 19 (CD19): B-lymphocytes, and cluster of differentiation 56 (CD56): assumed natural killer cells, were determined using flow cytometry.
Time Frame: Month 1, 3, 6, 12
Population: FAS: all randomized participants who received at least 1 dose of study medication. Here, N (Number of Participants Analyzed) signifies participants evaluable for this measure; and 'n' signifies those participants who were evaluable at given time point for each group, respectively.
Measure: Mean (Standard Deviation); unit: cells per microliter
Arm/Group | Cyclosporine | CP-690,550 15 mg for Months 1 to 6 | CP-690,550 15 mg for Months 1 to 3
Number analyzed (Participants) | 60 | 54 | 47
cells per microliter
  CD3: Month 1 (n=60,54,47) | 1555.0 (925.45) | 1256.7 (708.47) | 1327.2 (627.74)
  CD3: Month 3 (n=59,44,34) | 1273.2 (742.82) | 894.20 (527.87) | 1007.1 (447.91)
  CD3: Month 6 (n=47,34,31) | 1267.9 (693.20) | 811.74 (379.16) | 970.39 (410.28)
  CD3: Month 12 (n=45,29,26) | 1352.5 (647.60) | 796.76 (368.51) | 956.04 (522.08)
  CD19: Month 1 (n=60,54,47) | 280.58 (220.96) | 409.39 (339.45) | 416.70 (304.95)
  CD19: Month 3 (n=58,44,34) | 154.47 (208.07) | 189.41 (190.23) | 185.68 (139.24)
  CD19: Month 6 (n=47,34,31) | 125.26 (164.65) | 151.03 (129.52) | 173.10 (136.53)
  CD19: Month 12 (n=45,29,26) | 120.18 (117.14) | 180.03 (235.85) | 181.46 (141.45)
  CD56: Month 1 (n=60,54,47) | 166.47 (93.95) | 116.65 (110.62) | 112.23 (110.25)
  CD56: Month 3 (n=58,44,34) | 143.14 (86.42) | 86.86 (97.80) | 65.38 (38.91)
  CD56: Month 6 (n=47,34,31) | 170.23 (123.27) | 68.06 (63.85) | 65.00 (48.86)
  CD56: Month 12 (n=45,29,26) | 168.91 (122.80) | 96.00 (100.85) | 77.23 (57.74)

12. Secondary Outcome: Population Pharmacokinetics (PK)
Description: Data for this Outcome Measure are not reported here because the analysis population includes participants who were not enrolled in this study. ClinicalTrials.gov is designed for reporting results from only those participants who were enrolled in the study and described in the Participant Flow and Baseline Characteristics modules.
Time Frame: Pre-dose-2(P-2), Pre-dose(P), 0.5,1,2 hr post-dose(PD) on Day14, Month(M) 3; P,1,2 hr PD on M1; P, 0.5, 2, 4 hr PD on M6; P-2, P, 0.5 hr PD on M9, M12 as per randomization in CP-690,550 treated; P on M3 and P, 2, 4 hr PD on M6 in CsA treated participants
Reporting Status: Not Posted
Measure: Mean (Standard Deviation); unit: nanogram*hour per milliliter (ng*hr/mL)

13. Secondary Outcome: Glomerular Filtration Rate (GFR) by The Nankivell Equation
Description: GFR: an index of kidney function. GFR described the flow rate of filtered fluid through the kidney. GFR was measured directly or estimated using established formulas. GFR was calculated was estimated by creatinine clearance (CLcr) using Nankivell equation. CLcr by Nankivell equation= (6.7 per serum creatinine) plus (0.25*body weight) minus (0.5*serum urea) minus (100 per height square) plus (35 for male/25 for female). A normal GFR is >90 mL/min, although children and older people usually have a lower GFR. Lower values indicated poor kidney function. A GFR <15 mL/min indicated kidney failure.
Time Frame: Month 1, 3, 6, 9, 12
Population: FAS: all randomized participants who received at least 1 dose of study medication. Here, N (Number of Participants Analyzed) signifies participants evaluable for this measure. Missing data were imputed using Last Observation Carried Forward (LOCF).
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Cyclosporine | CP-690,550 15 mg for Months 1 to 6 | CP-690,550 15 mg for Months 1 to 3
Number analyzed (Participants) | 105 | 100 | 95
mL/min
  Month 1 | 65.85 (19.73) | 71.53 (17.72) | 73.66 (16.53)
  Month 3 | 65.80 (17.88) | 73.58 (18.46) | 72.91 (16.90)
  Month 6 | 66.75 (18.75) | 73.23 (18.26) | 74.49 (16.81)
  Month 9 | 66.85 (20.33) | 74.29 (18.23) | 74.22 (16.78)
  Month 12 | 66.88 (21.87) | 75.58 (18.54) | 75.41 (17.50)

14. Secondary Outcome: Glomerular Filtration Rate (GFR) by The Cockcroft-Gault Equation
Description: GFR: an index of kidney function. GFR described the flow rate of filtered fluid through the kidney. GFR was measured directly or estimated using established formulas. GFR was calculated using Cockcroft-Gault equation. GFR by Cockcroft-Gault equation= body weight*(140 minus age in years) divided by (72*serum creatinine). For females value obtained was multiplied by 0.85. A normal GFR is >90 mL/min, although children and older people usually have a lower GFR. Lower values indicated poor kidney function. A GFR <15 mL/min indicated kidney failure.
Time Frame: Month 1, 3, 6, 9, 12
Population: FAS: all randomized participants who received at least 1 dose of study medication. Here, N (Number of Participants Analyzed) signifies participants evaluable for this measure. Missing data were imputed using LOCF.
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Cyclosporine | CP-690,550 15 mg for Months 1 to 6 | CP-690,550 15 mg for Months 1 to 3
Number analyzed (Participants) | 105 | 100 | 95
mL/min
  Month 1 | 67.23 (23.84) | 71.12 (23.31) | 73.55 (20.62)
  Month 3 | 68.08 (23.19) | 74.41 (25.76) | 74.16 (22.45)
  Month 6 | 69.21 (23.66) | 74.71 (25.87) | 76.30 (23.11)
  Month 9 | 70.05 (25.15) | 76.41 (25.62) | 76.40 (24.20)
  Month 12 | 69.67 (25.64) | 78.41 (27.62) | 78.09 (24.69)

15. Secondary Outcome: Glomerular Filtration Rate (GFR) by The Modification of Diet in Renal Disease (MDRD) Equation
Description: GFR: an index of kidney function. GFR described the flow rate of filtered fluid through the kidney. GFR was calculated using MDRD equation. GFR by MDRD equation = 170 * (serum creatinine)^(-0.999) * (age in years)^(-0.176) * (0.762 if female) * (1.18 if black) * (blood urea nitrogen concentration)^(-0.170) * (serum albumin concentration)^(0.318).A normal GFR is >90 mL/min/1.73 square meter (m^2), although children and older people usually have a lower GFR. Lower values indicated poor kidney function. A GFR <15 mL/min/1.73 m^2 indicated kidney failure.
Time Frame: Month 1, 3, 6, 9, 12
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: mL/min/1.73 m^2
Arm/Group | Cyclosporine | CP-690,550 15 mg for Months 1 to 6 | CP-690,550 15 mg for Months 1 to 3
Number analyzed (Participants) | 105 | 100 | 95
mL/min/1.73 m^2
  Month 1 | 52.89 (20.05) | 59.93 (17.54) | 63.61 (21.00)
  Month 3 | 53.55 (18.83) | 62.20 (17.16) | 62.81 (20.04)
  Month 6 | 54.16 (19.21) | 61.84 (17.71) | 64.04 (19.63)
  Month 9 | 54.11 (20.45) | 62.98 (17.50) | 63.61 (18.82)
  Month 12 | 53.94 (21.36) | 64.25 (18.28) | 64.59 (20.35)

16. Secondary Outcome: Glomerular Filtration Rate (GFR) by The Abbreviated Modification of Diet in Renal Disease (MDRD) Equation
Description: GFR: an index of kidney function. GFR described the flow rate of filtered fluid through the kidney. GFR was measured directly or estimated using established formulas. GFR was calculated using abbreviated MDRD equation. GFR by abbreviated MDRD equation= 186 * (serum creatinine)^(-1.154) * (age in years)^(-0.203) * (0.742 if female) * (1.210 if black). A normal GFR is >90 mL/min/1.73 m^2, although children and older people usually have a lower GFR. Lower values indicated poor kidney function. A GFR <15 mL/min/1.73 m^2 indicated kidney failure.
Time Frame: Month 1, 3, 6, 9, 12
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: mL/min per 1.73 m^2
Arm/Group | Cyclosporine | CP-690,550 15 mg for Months 1 to 6 | CP-690,550 15 mg for Months 1 to 3
Number analyzed (Participants) | 105 | 100 | 95
mL/min per 1.73 m^2
  Month 1 | 55.29 (21.96) | 61.49 (18.66) | 64.81 (21.15)
  Month 3 | 54.36 (19.28) | 62.45 (18.39) | 62.27 (19.71)
  Month 6 | 55.01 (20.22) | 61.49 (18.10) | 63.33 (19.74)
  Month 9 | 55.39 (22.09) | 62.52 (17.86) | 62.76 (18.55)
  Month 12 | 54.99 (24.15) | 63.88 (18.40) | 64.17 (19.94)

17. Secondary Outcome: Number of Participants With Clinically Significant Infections
Description: Clinically significant infection was defined as the presence of documented infection confirmed by culture, biopsy, genomic, or serologic findings post-randomization and requiring hospitalization or parenteral anti-infective treatment, or otherwise deemed significant by the investigator.
Time Frame: Baseline up to Month 12
Population: FAS: all randomized participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | Cyclosporine | CP-690,550 15 mg for Months 1 to 6 | CP-690,550 15 mg for Months 1 to 3
Number analyzed (Participants) | 109 | 106 | 107
participants | 61 | 88 | 83

18. Secondary Outcome: 36-Item Short-Form Health Survey (SF-36)
Description: SF-36: standardized survey evaluating 8 aspects of functional health and well-being: physical and social functioning, physical and emotional role limitations, bodily pain, general health, vitality, mental health. These 8 aspects can also be summarized as physical and mental component scores. Total of 11 variables were analyzed (8 subscales,2 composite subscales and Question(Q) 2 "how would you rate your health in general now?"(range 1=better, 5=worst). The score for a section (except Q2) is an average of the individual question scores, which are scaled 0-100 (100=highest level of functioning).
Time Frame: Baseline, Month 6, 12
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cyclosporine | CP-690,550 15 mg for Months 1 to 6 | CP-690,550 15 mg for Months 1 to 3
Number analyzed (Participants) | 80 | 68 | 72
units on a scale
  Baseline: Bodily Pain (n=79,68,71) | 52.89 (9.45) | 51.43 (10.56) | 49.56 (10.59)
  Baseline: General Health (n=79,68,72) | 44.77 (9.28) | 42.46 (10.63) | 42.39 (9.68)
  Baseline: Mental Health (n=78,68,72) | 49.15 (9.13) | 44.85 (12.75) | 48.69 (11.33)
  Baseline: Physical Functioning (n=79,68,72) | 44.03 (10.03) | 44.46 (9.58) | 45.88 (9.52)
  Baseline: Role Emotional (n=79,68,71) | 46.19 (11.75) | 43.82 (13.80) | 43.79 (13.62)
  Baseline: Role Physical (n=79,68,71) | 41.26 (11.86) | 42.28 (12.56) | 42.51 (12.32)
  Baseline: Social Functioning (n=79,68,72) | 47.42 (8.98) | 41.14 (12.42) | 44.38 (11.54)
  Baseline: Vitality (n=78,68,72) | 49.77 (10.81) | 48.04 (12.38) | 50.29 (10.57)
  Baseline: Physical Component (n=78,68,71) | 44.85 (9.38) | 45.85 (8.35) | 45.05 (8.58)
  Baseline: Mental Component (n=78,68,71) | 49.41 (9.66) | 44.18 (13.27) | 47.13 (11.54)
  Baseline: Q2-Health in General Now (n=80,68,72) | 2.78 (0.62) | 2.57 (0.78) | 2.63 (0.74)
  Month 6: Bodily Pain (n=78,63,65) | 51.87 (9.55) | 49.76 (11.49) | 50.88 (10.10)
  Month 6: General Health (n=78,63,65) | 47.87 (9.00) | 46.70 (10.31) | 47.36 (9.79)
  Month 6: Mental Health (n=78,63,65) | 50.47 (10.69) | 48.35 (12.48) | 48.81 (10.97)
  Month 6: Physical Functioning (n=77,63,65) | 47.06 (9.96) | 45.74 (11.08) | 46.91 (10.50)
  Month 6: Role Emotional (n=77,63,65) | 48.06 (11.15) | 45.40 (11.82) | 46.77 (11.87)
  Month 6: Role Physical (n=77,63,65) | 46.48 (10.44) | 43.11 (12.14) | 45.87 (10.80)
  Month 6: Social Functioning (n=78,63,65) | 50.34 (8.64) | 45.14 (12.21) | 47.88 (10.15)
  Month 6: Vitality (n=78,63,65) | 54.22 (9.70) | 52.13 (11.14) | 51.95 (10.49)
  Month 6: Physical Component (n=77,63,65) | 47.93 (8.27) | 46.22 (10.76) | 47.82 (9.24)
  Month 6: Mental Component (n=77,63,65) | 51.60 (9.43) | 48.30 (11.82) | 49.09 (10.91)
  Month 6: Q2-Health in General Now (n=78,63,65) | 2.74 (0.73) | 2.65 (0.77) | 2.72 (0.63)
  Month 12: Bodily Pain (n=73,58,56) | 51.12 (9.23) | 51.07 (10.24) | 49.48 (10.95)
  Month 12: General Health (n=73,57,56) | 48.94 (8.74) | 46.79 (8.71) | 44.71 (10.02)
  Month 12: Mental Health (n=73,57,56) | 51.93 (9.24) | 49.43 (10.98) | 46.91 (10.77)
  Month 12: Physical Functioning (n=73,58,56) | 47.19 (10.26) | 46.88 (10.16) | 46.99 (11.01)
  Month 12: Role Emotional (n=71,57,56) | 46.13 (12.36) | 47.31 (9.15) | 46.21 (12.27)
  Month 12: Role Physical (n=71,57,56) | 46.57 (9.68) | 44.19 (10.73) | 45.20 (11.47)
  Month 12: Social Functioning (n=73,57,56) | 49.63 (8.41) | 46.87 (10.06) | 47.18 (10.84)
  Month 12: Vitality (n=73,57,56) | 54.25 (8.31) | 51.45 (11.20) | 51.69 (10.23)
  Month 12: Physical Component (n=71,57,56) | 47.98 (8.02) | 46.84 (8.80) | 47.03 (10.23)
  Month 12: Mental Component (n=71,57,56) | 51.12 (9.34) | 49.47 (9.36) | 47.91 (12.17)
  Month 12: Q2-Health in General Now (n=73,58,56) | 2.75 (0.62) | 2.69 (0.71) | 2.84 (0.56)

19. Secondary Outcome: End-Stage Renal Disease Symptom Checklist Transplantation Module (ESRD-SCL)
Description: ESRD-SCL:43-item disease specific self-administered questionnaire. Participants' rated question"At the moment,how much do you suffer?"for each item on 5 point scale,ranged (Ra) 0(not at all)to 4(extremely).Consisted of 6 subscales:cardiac and renal dysfunction;Ra 0-28,increased(In) growth of gum and hair;Ra 0-20,limited cognitive capacity;Ra 0-32,limited physical capacity;Ra 0 - 40,side effects (SEs) of corticosteroids;Ra 0-20,transplantation associated psychological distress(TAPD);Ra 0-32(higher scores=greater dysfunction for each subscale).Total score:0-172,higher scores=greater dysfunction.
Time Frame: Baseline, Month 6, 12
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cyclosporine | CP-690,550 15 mg for Months 1 to 6 | CP-690,550 15 mg for Months 1 to 3
Number analyzed (Participants) | 77 | 64 | 71
units on a scale
  Baseline:Cardiac and Renal Dysfunction(n=76,61,71) | 0.76 (0.55) | 0.70 (0.59) | 0.64 (0.61)
  Baseline: In Growth of Gum and Hair (n=76,61,70) | 0.19 (0.36) | 0.16 (0.31) | 0.18 (0.32)
  Baseline: Limited Cognitive Capacity (n=77,62,71) | 0.67 (0.63) | 0.76 (0.74) | 0.64 (0.61)
  Baseline: Limited Physical Capacity (n=76,61,71) | 0.80 (0.59) | 0.79 (0.65) | 0.72 (0.56)
  Baseline: SEs of Corticosteroids (n=76,61,71) | 0.45 (0.53) | 0.56 (0.64) | 0.48 (0.52)
  Baseline: TAPD (n=77,62,71) | 0.98 (0.68) | 1.21 (0.82) | 1.16 (0.74)
  Month 6:Cardiac and Renal Dysfunction(n=77,63,64) | 0.59 (0.63) | 0.40 (0.50) | 0.50 (0.48)
  Month 6: In Growth of Gum and Hair (n=77,63,64) | 0.67 (0.61) | 0.23 (0.47) | 0.24 (0.35)
  Month 6: Limited Cognitive Capacity (n=77,64,65) | 0.64 (0.68) | 0.70 (0.74) | 0.68 (0.50)
  Month 6: Limited Physical Capacity (n=77,63,64) | 0.69 (0.60) | 0.67 (0.61) | 0.62 (0.49)
  Month 6: SEs of Corticosteroids (n=77,63,64) | 0.65 (0.70) | 0.54 (0.56) | 0.69 (0.63)
  Month 6: TAPD (n=77,64,65) | 0.62 (0.60) | 0.78 (0.65) | 0.85 (0.62)
  Month 12:Cardiac and Renal Dysfunction(n=70,57,55) | 0.51 (0.46) | 0.51 (0.48) | 0.49 (0.50)
  Month 12: In Growth of Gum and Hair (n=70,57,55) | 0.58 (0.52) | 0.19 (0.30) | 0.29 (0.51)
  Month 12: Limited Cognitive Capacity (n=71,58,55) | 0.68 (0.60) | 0.79 (0.70) | 0.85 (0.67)
  Month 12: Limited Physical Capacity (n=70,57,55) | 0.63 (0.46) | 0.69 (0.50) | 0.73 (0.65)
  Month 12: SEs of Corticosteroids (n=70,56,55) | 0.50 (0.48) | 0.56 (0.63) | 0.72 (0.78)
  Month 12: TAPD (n=71,57,55) | 0.58 (0.53) | 0.90 (0.66) | 0.96 (0.73)

20. Secondary Outcome: Severity of Dyspepsia Assessment (SODA)
Description: SODA:17-item health scale, assessed participant-reported perceptions of dyspepsia;consists of 3 subscales:Pain Intensity (6-items to assess pain and intensity of abdominal [Ab] discomfort; Range (Ra):2-47, higher score= greater pain and Ab discomfort), Non-Pain Symptoms (7-items to assess severity and impact of non-pain symptoms:burping/belching,heartburn,bloating,flatulence,sour taste,nausea,and bad breath; Ra:7-35,higher scores = increased symptom severity and influence), and Satisfaction (4-items to assess degree of satisfaction with Ab discomfort; Ra:2-23,higher scores= more satisfaction).
Time Frame: Baseline, Month 6, 12
Population: Data not analyzed since the SODA instrument was found irrelevant in the treated population.
Arm/Group | Cyclosporine | CP-690,550 15 mg for Months 1 to 6 | CP-690,550 15 mg for Months 1 to 3
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Cyclosporine | CP-690,550 15 mg for Months 1 to 6 | CP-690,550 15 mg for Months 1 to 3
Serious Adverse Events (participants affected / at risk) | 65/109 | 76/106 | 74/107
Other Adverse Events (participants affected / at risk) | 105/109 | 102/106 | 105/107
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cyclosporine (N=109) | CP-690,550 15 mg for Months 1 to 6 (N=106) | CP-690,550 15 mg for Months 1 to 3 (N=107)
Anaemia (Blood and lymphatic system disorders) | 2 | 5 | 8
Aplastic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 6 | 2
Neutropenia (Blood and lymphatic system disorders) | 0 | 2 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 1
Angina unstable (Cardiac disorders) | 1 | 0 | 0
Arrhythmia (Cardiac disorders) | 0 | 1 | 0
Arrhythmia supraventricular (Cardiac disorders) | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 2 | 0
Atrial flutter (Cardiac disorders) | 0 | 0 | 1
Bradycardia (Cardiac disorders) | 1 | 0 | 0
Cardiac arrest (Cardiac disorders) | 1 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 1 | 0
Electromechanical dissociation (Cardiac disorders) | 0 | 0 | 1
Left ventricular hypertrophy (Cardiac disorders) | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1 | 2
Tachycardia (Cardiac disorders) | 0 | 0 | 1
Congenital cystic kidney disease (Congenital, familial and genetic disorders) | 0 | 0 | 1
Adrenal mass (Endocrine disorders) | 1 | 0 | 0
Blindness cortical (Eye disorders) | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 3 | 2
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 1 | 0
Colitis ischaemic (Gastrointestinal disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 4 | 1
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 0 | 1 | 0
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 0
Intestinal perforation (Gastrointestinal disorders) | 1 | 0 | 0
Large intestine perforation (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 0 | 2
Pancreatitis necrotising (Gastrointestinal disorders) | 1 | 0 | 0
Peritonitis (Gastrointestinal disorders) | 1 | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Reflux oesophagitis (Gastrointestinal disorders) | 0 | 1 | 0
Retroperitoneal haematoma (Gastrointestinal disorders) | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 3 | 2 | 1
Brain death (General disorders) | 0 | 2 | 0
Chills (General disorders) | 1 | 0 | 0
Condition aggravated (General disorders) | 0 | 1 | 0
Drug interaction (General disorders) | 0 | 1 | 1
Hernia (General disorders) | 0 | 1 | 0
Multi-organ failure (General disorders) | 1 | 0 | 0
Oedema peripheral (General disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 2 | 5 | 4
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0 | 0
Kidney transplant rejection (Immune system disorders) | 8 | 5 | 5
Serum sickness (Immune system disorders) | 0 | 1 | 0
Transplant rejection (Immune system disorders) | 9 | 14 | 10
Abdominal abscess (Infections and infestations) | 0 | 0 | 1
Acute sinusitis (Infections and infestations) | 0 | 0 | 1
Appendicitis (Infections and infestations) | 1 | 0 | 0
Arteriovenous fistula site infection (Infections and infestations) | 0 | 1 | 0
BK virus infection (Infections and infestations) | 0 | 1 | 4
Bacteraemia (Infections and infestations) | 3 | 0 | 1
Bacterial pyelonephritis (Infections and infestations) | 0 | 1 | 0
Bacterial sepsis (Infections and infestations) | 0 | 0 | 1
Bacteriuria (Infections and infestations) | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1
Bronchopulmonary aspergillosis (Infections and infestations) | 0 | 1 | 1
Cellulitis (Infections and infestations) | 0 | 1 | 0
Cystitis (Infections and infestations) | 0 | 0 | 1
Cytomegalovirus colitis (Infections and infestations) | 0 | 1 | 1
Cytomegalovirus gastroenteritis (Infections and infestations) | 0 | 0 | 1
Cytomegalovirus infection (Infections and infestations) | 2 | 10 | 7
Cytomegalovirus oesophagitis (Infections and infestations) | 0 | 1 | 0
Cytomegalovirus viraemia (Infections and infestations) | 1 | 10 | 1
Diarrhoea infectious (Infections and infestations) | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 1 | 0
Enterococcal bacteraemia (Infections and infestations) | 0 | 0 | 1
Escherichia urinary tract infection (Infections and infestations) | 1 | 0 | 0
Gangrene (Infections and infestations) | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 2
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 1
Genital herpes (Infections and infestations) | 0 | 0 | 1
Haematoma infection (Infections and infestations) | 1 | 0 | 0
Herpes ophthalmic (Infections and infestations) | 1 | 0 | 0
Herpes virus infection (Infections and infestations) | 0 | 1 | 1
Herpes zoster (Infections and infestations) | 1 | 3 | 1
Incision site infection (Infections and infestations) | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 0 | 1
Keratitis herpetic (Infections and infestations) | 1 | 0 | 0
Klebsiella bacteraemia (Infections and infestations) | 0 | 1 | 0
Klebsiella sepsis (Infections and infestations) | 0 | 1 | 0
Localised infection (Infections and infestations) | 0 | 1 | 0
Lung infection (Infections and infestations) | 0 | 1 | 1
Oral herpes (Infections and infestations) | 0 | 1 | 0
Osteomyelitis (Infections and infestations) | 0 | 1 | 1
Perinephric abscess (Infections and infestations) | 1 | 0 | 0
Peritoneal infection (Infections and infestations) | 0 | 1 | 0
Pneumocystis jiroveci pneumonia (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 4 | 2 | 1
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 | 0 | 1
Polyomavirus-associated nephropathy (Infections and infestations) | 0 | 0 | 2
Postoperative wound infection (Infections and infestations) | 0 | 0 | 1
Prostatic abscess (Infections and infestations) | 0 | 0 | 1
Pseudomonas infection (Infections and infestations) | 0 | 0 | 1
Pyelonephritis (Infections and infestations) | 2 | 2 | 1
Pyelonephritis acute (Infections and infestations) | 1 | 0 | 1
Retinitis viral (Infections and infestations) | 0 | 1 | 1
Sepsis (Infections and infestations) | 1 | 3 | 2
Septic shock (Infections and infestations) | 1 | 2 | 1
Staphylococcal bacteraemia (Infections and infestations) | 0 | 0 | 1
Tuberculosis (Infections and infestations) | 1 | 0 | 0
Tuberculosis gastrointestinal (Infections and infestations) | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 0
Urinary tract infection (Infections and infestations) | 6 | 11 | 5
Urinary tract infection bacterial (Infections and infestations) | 1 | 0 | 0
Urinary tract infection enterococcal (Infections and infestations) | 1 | 0 | 0
Urinary tract infection fungal (Infections and infestations) | 0 | 1 | 0
Urosepsis (Infections and infestations) | 1 | 0 | 0
Viral infection (Infections and infestations) | 1 | 0 | 0
Wound infection (Infections and infestations) | 0 | 2 | 2
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1 | 0
Anaemia postoperative (Injury, poisoning and procedural complications) | 1 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 1 | 0 | 0
Chronic allograft nephropathy (Injury, poisoning and procedural complications) | 1 | 0 | 0
Complications of transplanted kidney (Injury, poisoning and procedural complications) | 0 | 1 | 0
Compression fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Graft complication (Injury, poisoning and procedural complications) | 0 | 6 | 5
Graft dysfunction (Injury, poisoning and procedural complications) | 3 | 2 | 0
Graft loss (Injury, poisoning and procedural complications) | 1 | 0 | 0
Graft thrombosis (Injury, poisoning and procedural complications) | 0 | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1
Patella fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Perirenal haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1
Post procedural discharge (Injury, poisoning and procedural complications) | 1 | 0 | 0
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1
Post procedural haematuria (Injury, poisoning and procedural complications) | 1 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 2 | 0 | 0
Postoperative wound complication (Injury, poisoning and procedural complications) | 0 | 1 | 0
Renal graft loss (Injury, poisoning and procedural complications) | 0 | 1 | 0
Renal lymphocele (Injury, poisoning and procedural complications) | 0 | 0 | 1
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0
Urethral injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 | 1 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 2 | 1 | 4
Wound secretion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Blood creatine increased (Investigations) | 0 | 1 | 0
Blood creatinine increased (Investigations) | 9 | 7 | 6
Blood pressure increased (Investigations) | 0 | 1 | 0
Blood urea increased (Investigations) | 1 | 0 | 0
Electroencephalogram abnormal (Investigations) | 0 | 1 | 0
Hepatic enzyme increased (Investigations) | 0 | 1 | 0
Liver function test abnormal (Investigations) | 0 | 1 | 0
Transaminases increased (Investigations) | 0 | 0 | 1
Troponin I increased (Investigations) | 0 | 1 | 0
White blood cell count increased (Investigations) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 2
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 2 | 0 | 0
Fluid overload (Metabolism and nutrition disorders) | 1 | 1 | 0
Hypercreatininaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 3 | 2 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Myopathy (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Epstein-Barr virus associated lymphoproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Areflexia (Nervous system disorders) | 0 | 1 | 0
Brain oedema (Nervous system disorders) | 0 | 1 | 0
Cerebral infarction (Nervous system disorders) | 1 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 2 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 1
Embolic stroke (Nervous system disorders) | 0 | 1 | 0
Encephalopathy (Nervous system disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 1
Intracranial pressure increased (Nervous system disorders) | 0 | 1 | 0
Loss of consciousness (Nervous system disorders) | 0 | 0 | 1
Sciatica (Nervous system disorders) | 1 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 2 | 0
Bladder irritation (Renal and urinary disorders) | 1 | 0 | 0
Bladder spasm (Renal and urinary disorders) | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 1 | 2 | 3
Haemorrhage urinary tract (Renal and urinary disorders) | 0 | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 2 | 1 | 0
Nephropathy toxic (Renal and urinary disorders) | 1 | 0 | 1
Polyuria (Renal and urinary disorders) | 0 | 1 | 0
Renal artery occlusion (Renal and urinary disorders) | 0 | 0 | 1
Renal artery stenosis (Renal and urinary disorders) | 2 | 0 | 0
Renal cyst (Renal and urinary disorders) | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 2 | 5 | 0
Renal impairment (Renal and urinary disorders) | 1 | 1 | 0
Renal tubular necrosis (Renal and urinary disorders) | 1 | 1 | 2
Renal vein thrombosis (Renal and urinary disorders) | 0 | 0 | 1
Ureteric obstruction (Renal and urinary disorders) | 1 | 0 | 1
Urethral stenosis (Renal and urinary disorders) | 0 | 1 | 0
Urinary fistula (Renal and urinary disorders) | 1 | 0 | 2
Urinary incontinence (Renal and urinary disorders) | 1 | 2 | 0
Urinary retention (Renal and urinary disorders) | 2 | 3 | 1
Urinary tract obstruction (Renal and urinary disorders) | 0 | 1 | 0
Epididymitis (Reproductive system and breast disorders) | 1 | 0 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Bladder catheter removal (Surgical and medical procedures) | 1 | 0 | 0
Arterial haemorrhage (Vascular disorders) | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 3 | 1
Haematoma (Vascular disorders) | 0 | 1 | 1
Haemorrhage (Vascular disorders) | 0 | 0 | 1
Hypertension (Vascular disorders) | 2 | 1 | 0
Hypotension (Vascular disorders) | 1 | 1 | 0
Ischaemia (Vascular disorders) | 0 | 1 | 0
Lymphocele (Vascular disorders) | 1 | 2 | 3
Malignant hypertension (Vascular disorders) | 1 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 1
Superior vena caval occlusion (Vascular disorders) | 0 | 0 | 1
Thrombosis (Vascular disorders) | 1 | 0 | 0
Vascular insufficiency (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cyclosporine (N=109) | CP-690,550 15 mg for Months 1 to 6 (N=106) | CP-690,550 15 mg for Months 1 to 3 (N=107)
Anaemia (Blood and lymphatic system disorders) | 26 | 46 | 38
Leukocytosis (Blood and lymphatic system disorders) | 0 | 3 | 4
Leukopenia (Blood and lymphatic system disorders) | 12 | 26 | 17
Lymphopenia (Blood and lymphatic system disorders) | 2 | 2 | 3
Neutropenia (Blood and lymphatic system disorders) | 2 | 12 | 4
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1 | 3
Polycythaemia (Blood and lymphatic system disorders) | 3 | 3 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 1 | 4
Thrombocytosis (Blood and lymphatic system disorders) | 1 | 3 | 0
Bradycardia (Cardiac disorders) | 3 | 3 | 1
Left ventricular hypertrophy (Cardiac disorders) | 1 | 3 | 0
Palpitations (Cardiac disorders) | 2 | 4 | 1
Sinus tachycardia (Cardiac disorders) | 3 | 2 | 2
Tachycardia (Cardiac disorders) | 3 | 7 | 8
Vision blurred (Eye disorders) | 1 | 3 | 1
Visual impairment (Eye disorders) | 3 | 3 | 1
Abdominal discomfort (Gastrointestinal disorders) | 2 | 4 | 3
Abdominal distension (Gastrointestinal disorders) | 10 | 6 | 8
Abdominal pain (Gastrointestinal disorders) | 15 | 15 | 4
Abdominal pain upper (Gastrointestinal disorders) | 6 | 6 | 2
Aphthous stomatitis (Gastrointestinal disorders) | 2 | 4 | 0
Ascites (Gastrointestinal disorders) | 1 | 1 | 4
Constipation (Gastrointestinal disorders) | 30 | 35 | 38
Diarrhoea (Gastrointestinal disorders) | 22 | 26 | 29
Dyspepsia (Gastrointestinal disorders) | 6 | 8 | 5
Flatulence (Gastrointestinal disorders) | 1 | 3 | 2
Gastritis (Gastrointestinal disorders) | 0 | 2 | 3
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 3 | 4
Gingival hypertrophy (Gastrointestinal disorders) | 4 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 2 | 5 | 0
Hiatus hernia (Gastrointestinal disorders) | 0 | 3 | 0
Mouth ulceration (Gastrointestinal disorders) | 1 | 0 | 3
Nausea (Gastrointestinal disorders) | 23 | 29 | 25
Vomiting (Gastrointestinal disorders) | 18 | 15 | 12
Asthenia (General disorders) | 2 | 4 | 3
Chest pain (General disorders) | 3 | 4 | 3
Chills (General disorders) | 3 | 1 | 2
Fatigue (General disorders) | 11 | 9 | 15
Influenza like illness (General disorders) | 3 | 1 | 2
Oedema (General disorders) | 12 | 15 | 11
Oedema peripheral (General disorders) | 30 | 25 | 19
Pain (General disorders) | 2 | 3 | 1
Pyrexia (General disorders) | 12 | 16 | 15
Transplant rejection (Immune system disorders) | 14 | 8 | 5
BK virus infection (Infections and infestations) | 6 | 14 | 15
Bronchitis (Infections and infestations) | 2 | 4 | 3
Candidiasis (Infections and infestations) | 3 | 0 | 1
Cytomegalovirus infection (Infections and infestations) | 1 | 4 | 2
Cytomegalovirus viraemia (Infections and infestations) | 12 | 21 | 18
Epstein-Barr viraemia (Infections and infestations) | 0 | 3 | 2
Folliculitis (Infections and infestations) | 0 | 0 | 3
Fungal skin infection (Infections and infestations) | 0 | 3 | 1
Gastroenteritis (Infections and infestations) | 4 | 1 | 0
Genital herpes (Infections and infestations) | 0 | 3 | 2
Herpes simplex (Infections and infestations) | 3 | 2 | 3
Herpes zoster (Infections and infestations) | 3 | 5 | 6
Nasopharyngitis (Infections and infestations) | 4 | 7 | 7
Oral candidiasis (Infections and infestations) | 3 | 7 | 7
Oral herpes (Infections and infestations) | 0 | 4 | 5
Pneumonia (Infections and infestations) | 1 | 3 | 1
Polyomavirus-associated nephropathy (Infections and infestations) | 1 | 3 | 2
Rhinitis (Infections and infestations) | 1 | 3 | 0
Sinusitis (Infections and infestations) | 0 | 2 | 4
Upper respiratory tract infection (Infections and infestations) | 16 | 17 | 9
Urinary tract infection (Infections and infestations) | 25 | 19 | 22
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 3 | 2 | 1
Complications of transplant surgery (Injury, poisoning and procedural complications) | 3 | 2 | 6
Complications of transplanted kidney (Injury, poisoning and procedural complications) | 1 | 3 | 2
Contusion (Injury, poisoning and procedural complications) | 0 | 2 | 3
Foot fracture (Injury, poisoning and procedural complications) | 0 | 4 | 1
Graft complication (Injury, poisoning and procedural complications) | 10 | 7 | 14
Incision site pain (Injury, poisoning and procedural complications) | 3 | 9 | 11
Post procedural discharge (Injury, poisoning and procedural complications) | 4 | 1 | 4
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 | 1 | 3
Procedural hypotension (Injury, poisoning and procedural complications) | 3 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 14 | 21 | 15
Wound complication (Injury, poisoning and procedural complications) | 1 | 3 | 4
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 5 | 4
Wound secretion (Injury, poisoning and procedural complications) | 2 | 7 | 2
Alanine aminotransferase increased (Investigations) | 0 | 2 | 4
Blood creatine phosphokinase increased (Investigations) | 0 | 3 | 2
Blood creatinine increased (Investigations) | 12 | 11 | 15
Cardiac murmur (Investigations) | 3 | 5 | 2
Hepatic enzyme increased (Investigations) | 1 | 2 | 4
Liver function test abnormal (Investigations) | 2 | 5 | 2
Urine output decreased (Investigations) | 2 | 2 | 3
Viral test positive (Investigations) | 5 | 5 | 3
Weight decreased (Investigations) | 0 | 2 | 4
Weight increased (Investigations) | 14 | 15 | 12
White blood cell count decreased (Investigations) | 3 | 1 | 1
White blood cell count increased (Investigations) | 1 | 3 | 0
Acidosis (Metabolism and nutrition disorders) | 2 | 3 | 1
Decreased appetite (Metabolism and nutrition disorders) | 3 | 5 | 3
Dehydration (Metabolism and nutrition disorders) | 4 | 5 | 3
Diabetes mellitus (Metabolism and nutrition disorders) | 6 | 5 | 4
Dyslipidaemia (Metabolism and nutrition disorders) | 5 | 7 | 6
Fluid overload (Metabolism and nutrition disorders) | 5 | 11 | 5
Glucose tolerance impaired (Metabolism and nutrition disorders) | 3 | 3 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 10 | 4 | 6
Hypercholesterolaemia (Metabolism and nutrition disorders) | 5 | 10 | 8
Hyperglycaemia (Metabolism and nutrition disorders) | 13 | 10 | 7
Hyperkalaemia (Metabolism and nutrition disorders) | 12 | 16 | 18
Hyperlipidaemia (Metabolism and nutrition disorders) | 13 | 10 | 10
Hyperphosphataemia (Metabolism and nutrition disorders) | 2 | 2 | 3
Hypocalcaemia (Metabolism and nutrition disorders) | 4 | 12 | 4
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 3 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 13 | 11
Hypomagnesaemia (Metabolism and nutrition disorders) | 8 | 2 | 6
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 2 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 13 | 14 | 10
Metabolic acidosis (Metabolism and nutrition disorders) | 2 | 3 | 5
Vitamin D deficiency (Metabolism and nutrition disorders) | 2 | 0 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 9 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 7 | 11
Muscle spasms (Musculoskeletal and connective tissue disorders) | 5 | 5 | 8
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 5 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 9 | 5
Dizziness (Nervous system disorders) | 9 | 9 | 9
Headache (Nervous system disorders) | 14 | 13 | 20
Hypoaesthesia (Nervous system disorders) | 2 | 7 | 3
Lethargy (Nervous system disorders) | 2 | 1 | 4
Paraesthesia (Nervous system disorders) | 3 | 3 | 2
Sensory disturbance (Nervous system disorders) | 0 | 0 | 3
Tremor (Nervous system disorders) | 19 | 8 | 8
Anxiety (Psychiatric disorders) | 3 | 5 | 6
Depression (Psychiatric disorders) | 3 | 3 | 4
Insomnia (Psychiatric disorders) | 13 | 6 | 10
Bladder spasm (Renal and urinary disorders) | 3 | 2 | 1
Dysuria (Renal and urinary disorders) | 8 | 13 | 8
Haematuria (Renal and urinary disorders) | 10 | 15 | 9
Hydronephrosis (Renal and urinary disorders) | 3 | 6 | 4
Nephropathy toxic (Renal and urinary disorders) | 3 | 0 | 0
Nocturia (Renal and urinary disorders) | 1 | 4 | 1
Pollakiuria (Renal and urinary disorders) | 3 | 3 | 5
Polyuria (Renal and urinary disorders) | 1 | 3 | 2
Proteinuria (Renal and urinary disorders) | 9 | 4 | 6
Renal artery stenosis (Renal and urinary disorders) | 1 | 2 | 3
Renal impairment (Renal and urinary disorders) | 2 | 5 | 1
Renal tubular necrosis (Renal and urinary disorders) | 2 | 6 | 3
Urinary incontinence (Renal and urinary disorders) | 1 | 4 | 3
Urinary retention (Renal and urinary disorders) | 0 | 4 | 2
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 3 | 2
Penile pain (Reproductive system and breast disorders) | 4 | 2 | 2
Testicular swelling (Reproductive system and breast disorders) | 0 | 0 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 16 | 7
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 | 11 | 8
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 2
Rales (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 6 | 1 | 1
Acne (Skin and subcutaneous tissue disorders) | 4 | 14 | 18
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 5 | 5
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 3 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 4 | 4 | 4
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 3
Hirsutism (Skin and subcutaneous tissue disorders) | 9 | 1 | 0
Hypertrichosis (Skin and subcutaneous tissue disorders) | 5 | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 2 | 4 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 5 | 0
Rash (Skin and subcutaneous tissue disorders) | 7 | 12 | 6
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 3 | 2
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 4
Incisional drainage (Surgical and medical procedures) | 0 | 3 | 0
Deep vein thrombosis (Vascular disorders) | 3 | 3 | 1
Haematoma (Vascular disorders) | 1 | 5 | 0
Hypertension (Vascular disorders) | 30 | 24 | 23
Hypotension (Vascular disorders) | 6 | 18 | 13
Lymphocele (Vascular disorders) | 3 | 5 | 1
Orthostatic hypotension (Vascular disorders) | 1 | 5 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.